CLINICAL TRIAL: NCT06373354
Title: Comparison of Conspicuity of Masses and Architectural Distortions Between Wide- and Narrow-angle Digital Breast Tomosynthesis Systems
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Siemens Medical Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-0924; NCI-2024-03341 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Architectural Distortions; Breast Tomosynthesis
MeSH Terms: interventions — Mammography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Digital Breast Tomosynthesis (DBT): Participants that agree to take part in this study, your standard follow-up imaging will be done using an FDA approved DBT system, but it will be different from the DBT system used for your routine screening. For example, if narrow-angle DBT was used for your routine screening, then you will have standard wide-angle DBT. If wide-angle DBT used for your routine screening, then you will have narrow-angle DBT. These images will be used for diagnosis and to help decide your further care.
  Interventions: Device: Digital Breast Tomosynthesis (DBT)

INTERVENTIONS:
Device: Digital Breast Tomosynthesis (DBT) — Undergo tomosynthesis imaging

SUMMARY:
To compare narrow-angle digital breast tomosynthesis (DBT) and wide-angle DBT.

DETAILED DESCRIPTION:
Primary Objectives

- The primary objective of this proposed study is to show that bWBT (B.brilliant wide-angle breast tomosynthesis) images provide better lesion conspicuity for masses and architectural distortions than NBT images based on the standard screening tomosynthesis imaging.

Secondary Objectives

* The secondary objective of this proposed study is to show that WBT images provide better lesion conspicuity for masses and architectural distortions based on the standard screening tomosynthesis imaging.
* Additional secondary objectives include radiologist feedback on the B.brilliant images, technologist experience with B.brilliant, and a participant comfort survey.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing standard screening mammography.
* Ability to understand and sign consent.

Exclusion Criteria:

* Pregnant women.
* Women unable to consent.
* Male patients.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Screening mammography population at MD Anderson
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  ncidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Adrada, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org